CLINICAL TRIAL: NCT07388290
Title: The Effect of Centralization on Medial Meniscal Extrusion for Medial Meniscus Posterior Root Tear Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron Krych, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-011455
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Meniscus Tear
Keywords: Meniscus tear; Meniscus extrusion; Medial meniscus root repair; Meniscus centralization
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repair with meniscus centralization (Experimental): Medial meniscus posterior root tear (MMPRT) surgical repair with meniscus centralization
  Interventions: Procedure: Medial meniscus posterior root tear (MMPRT) repair with meniscus centralization
- Repair without centralization (Active Comparator): Medial meniscus posterior root tear (MMPRT) surgical repair without centralization
  Interventions: Procedure: Medial meniscus posterior root tear (MMPRT) repair without meniscus centralization

INTERVENTIONS:
Procedure: Medial meniscus posterior root tear (MMPRT) repair with meniscus centralization — The centralization technique involves placement of 1.8-mm Knotless FiberTak suture anchors along the periphery of the tibial plateau, starting from the posteromedial corner and progressing anteriorly. The anchors are deployed using a curved drill guide, and sutures are passed in a mattress configuration to re-tension the meniscotibial ligament to centralize the meniscus.
  Once centralization is complete, the posterior root tear is repaired using an anatomic suture anchor for aperture medial meniscus root fixation.
  Arms: Repair with meniscus centralization
Procedure: Medial meniscus posterior root tear (MMPRT) repair without meniscus centralization — The posterior root tear is repaired using an anatomic suture anchor for aperture medial meniscus root fixation.
  Arms: Repair without centralization

SUMMARY:
The purpose of this research is to determine if meniscus root repair with or without centralization will have an impact on postoperative pain, function, activity levels, patient satisfaction, and incidence of revision meniscus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Medial Meniscus Posterior Root Tear demonstrated on MRI
* Notable extrusion (>3 mm) on preoperative MRI
* Patient able to consent for themselves
* Patient agrees to comply with trial schedules and plan

Pre-operative Exclusion:

* Concomitant ligamentous or meniscal procedures
* Meniscal extrusion > 6 mm on pre-operative MRI
* Kellgren-Lawrence grade > 2
* Varus malalignment > 10 degrees
* Asymmetric varus alignment > 5 degrees
* Varus thrust while weightbearing
* Grade 3 bipolar medial compartment changes (isolated grade 3 changes on single articular surface with ≤ grade 2 changes on the opposing surface remains eligible)
* Previous surgery of the affected knee
* Associated fractures requiring surgery
* Concurrent Vascular injuries
* Hypermobility/Ehlers-Danlos Syndrome
* Inflammatory or autoimmune disease
* Severe mental/physical disability precluding post operative rehabilitation demands
* Contraindications to MRI
* Pregnant women

Arthroscopy Inclusion Criteria:

* Complete radial tears within 9 mm of medial meniscus posterior root
* ICRS Grade 3 or better

Arthroscopy Exclusion Criteria:

* Requiring concomitant procedures other than MMPRT
* ICRS Grade 4 changes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Meniscus extrusion measurement | Baseline (Preoperatively), 6 months
  Meniscus extrusion is measured in millimeters (mm) on coronal MRI at the level of the tibial spine

SECONDARY OUTCOMES:
Change in Kellgren-Lawrence grade on X-ray | Baseline (Screening), 12 months, 24 months
  The Kellgren-Lawrence (KL) system is a 0-4 scale used to grade the severity of knee osteoarthritis (OA) based on X-ray. It ranges from Grade 0 (no changes) to Grade 4 (severe).
Change in Tegner Activity Score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The Tegner Activity Questionnaire is a 1-item questionnaire rating physical activity from 0 (Disabled) to 10 (Elite competitive athlete). Total scores range from 0 - 10, with higher scores indicating a higher level of activity.
Change in Visual Analog Scale (VAS) Questionnaire score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The VAS is a 2-item questionnaire assessing pain using a scale of 0 (No pain) to 10 (Worst pain). Total scores range from 0 - 10, lower scores indicating lower pain and higher scores indicating greater pain.
Change in Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS, JR) Questionnaire score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The KOOS JR is a questionnaire designed to measure outcomes for patients with knee replacements. Questions focus on knee stiffness, pain, and function for daily activities and are assessed on a 5 point Likert-scale between 0 (None) and 4 (Extreme). Total scores range from 0 - 28, with higher scores indicating a greater impact of pain on daily functioning.
Change in International Knee Documentation Committee (IKDC) Questionnaire score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The International Knee Documentation Committee (IKDC) Subjective Knee Evaluation assesses overall function over 3 domains: symptoms, athletic activity, and knee function. Higher scores indicate higher levels of function and lower levels of symptoms.
Change in Likert Knee Questionnaire score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The Likert Knee Questionnaire is a 1-item survey asking the patient to rate knee pain post-surgery on a Likert scale where 0 (Much better than before surgery) and 5 (Much worse than before surgery).
Surgery Satisfaction Questionnaire | 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months
  The Surgery Satisfaction Questionnaire is a 1-item survey asking the patient to rate satisfaction with knee surgery on a Likert scale where 0 (Not at all) and 10 (Most Satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J. Krych, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - The Steadman Clinic, West Vail, Colorado
  - Hospital for Special Surgery at Naples Comprehensive Health (HSS at NCH),, Naples, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No